CLINICAL TRIAL: NCT01309763
Title: A Randomized, Controlled, Parallel Group, Patient-blinded, Single-center, Phase I Pilot Study to Assess the Tolerability and Safety of Repeated Administrations of a Single-dose of AFFITOPE AD03 to Alzheimer's Disease Patients
Brief Title: Safety and Tolerability of AFFITOPE AD03
Acronym: MimoVax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFF005A
Record Dates: First submitted 2009-09-02; First posted 2011-03-07 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — aluminum sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AFFITOPE AD03 (Active Comparator): s.c. injection
  Interventions: Biological: AFFITOPE AD03
- AFFITOPE AD03 + Alum (Experimental): s.c. injection
  Interventions: Biological: AFFITOPE AD03 + Alum

INTERVENTIONS:
Biological: AFFITOPE AD03 — s.c. injection
  Arms: AFFITOPE AD03
Biological: AFFITOPE AD03 + Alum — s.c. injection
  Arms: AFFITOPE AD03 + Alum

SUMMARY:
This is a randomized, controlled, parallel group, patient-blinded, single-center, phase I pilot study to assess tolerability and safety of repeated subcutaneous administration of a single-dose of AFFITOPE AD03 applied with or without adjuvant to patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease based on the NINCDS/ADRDA criteria.
* Assessing the severity of AD by the Mini Mental State Examination (MMSE). AD of mild degree has been confirmed if the MMSE score is in the range of 20 to 26.
* Hachinski Ischemia Scale is used to try and distinguish AD from multi-infarct dementia. A score of ≤ 4 suggests AD.
* The result of the Magnetic Resonance Imaging scan (MRI) of the patient's brain has to be consistent with the diagnosis of AD
* Written informed consent signed and dated by the patient and the caregiver. The patient's capability to give informed consent has to be confirmed by an independent psychiatrist or neurologist.
* Age between 50 and 80 years.
* Availability of a partner/caregiver knowing the patient and being able to accompany the patient at the visits and being available for the telephone interviews. This is necessary because some of the neuropsychiatric tests require information by a person knowing the patient well. In addition, it increases the safety of a study participant.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method.
* Availability of the APOE status
* A potential participant receiving conventional AD and hypothyroidism therapies must be on stable doses for at least 3 months prior to Visit 1 and during the entire trial period.
* A potential participant has to be on stable doses of all medications he/she is taking because of consisting illnesses according to medical history (except AD and hypothyroidism therapy itself which will be recorded separately) for at least 30 days prior to Visit 1, if considered relevant by the investigator.

Exclusion Criteria:

* Pregnant women.
* Sexually active women of childbearing potential who are not using a medically accepted birth control method.
* Participation in another clinical trial within 3 months before Visit 1.
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial.
* Presence or history of allergy to components of the vaccine, if considered relevant by the investigator.
* Contraindication for MRI imaging such as metallic endoprosthesis or stent implantation in the last 6 months or allergy to MRI contrast agent.
* Operation (under general anaesthesia) within 3 months prior to study entry and scheduled elective operation during the whole study period.
* History and/or presence of autoimmune disease, if considered relevant by the investigator.
* Recent (≤3 years since last specific treatment) history of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia).
* Active infectious disease (e.g., Hepatitis B, C).
* Presence and/or history of Immunodeficiency (e.g., HIV infection).
* Significant systemic illness (e.g., chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, other deficiencies), if considered relevant by the investigator.
* Hypothyroidism, defined as any significant thyroid-stimulating hormone elevation. Patients with corrected hypothyroidism are eligible for the study provided that treatment has been stable for 3 months before study entry.
* History of significant psychiatric illness such as schizophrenia, bipolar affective disorder or psychotic depression.
* Current depressive episode (Geriatric Depression Score (GDS) >5 at visit 1)
* Metabolic or toxic encephalopathy or dementia due to a general medical condition.
* Alcoholism or substance abuse within the past year (alcohol or drug intoxication).
* Wernicke's encephalopathy
* History or evidence of any other CNS disorder that could be interpreted as a cause of dementia (infectious or inflammatory/demyelinating CNS conditions, Creutzfeldt Jacob disease, Parkinson's disease, Huntington's disease, brain tumor, subdural haematoma, etc.)
* History or evidence of cerebrovascular disease (stroke, transient ischemic attack, hemorrhage), or diagnosis of possible, probable or definite vascular dementia in accordance with NINDS-AIREN criteria.
* Epilepsy
* Prior and/or current treatment with experimental immunotherapeutics including IVIG or vaccines for AD.
* Prior and/or current treatment with immunosuppressive drugs.
* Change in dose of standard treatments for AD or hypothyroidism within 3 months prior to visit 1.
* Change in dose of previous and current medications which the patient is taking because of consisting illnesses according medical history (except AD and hypothyroidism therapies, AD therapies will be recorded separately) within the last 30 days prior to visit 1, if clinically relevant.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
change in ADAS-Cog score as a measure of cognition | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, MD, Principal Investigator — MUW
Locations (1):
- MUW Wien, Vienna, Austria